CLINICAL TRIAL: NCT06723431
Title: Assessment of Pre Hospital Rescue Intervention for Seizure in Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Gamal Hussien, Assessment of pre hospital rescue intervention for seizure in pediatric patients, Assiut University
Other Study IDs: Pre hospital TTT of seizure
Record Dates: First submitted 2024-10-01; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Seizure
Keywords: seizure in pediatric patients
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- (A)Patient with seizure received rescue interventional (B) Patient with seizure didn't receive it: We will do 2 groups :
  Group A: Patient with recurrent attack of seizure and with prolonged seizure with prescribed treatment at home, Patients aged from 2 years to 18 years, Received rescue intervention.
  Group B: Patient with recurrent attack of seizure and with prolonged seizure without prescribed treatment at home, Patients aged from 2 years to 18 years, didn't Received rescue intervention.

SUMMARY:
1. Evaluation of pre hospital rescue intervention of seizure management.
2. To investigate the type of rescue medication, Efficacy, route of administration, Side effects of this drug, frequency and Indication of its use.

DETAILED DESCRIPTION:
An epileptic seizure is a transient occurrence with signs or symptoms due to abnormal excessive and synchronous neuronal activity in the brain.

There are many different types of seizures:

Current classification designates two large categories - partial or generalized. In a partial seizure, one area of the cortex is thought to be activated initially and may show simple symptoms such as a motor or sensory phenomena.

Partial seizures may rapidly secondarily generalize and spread to involve all cortical areas.

Generalized seizures result from diffuse cortical activation at seizure onset . Seizure cluster provides an opportunity to administer prompt treatment.

Delays in the treatment of seizure emergencies are often associated with negative patient outcomes.

Seizure clusters become less responsive to treatment when they continue unabated over time .

In addition to using anti epileptic medications, the treatment of seizures aims at correcting any identifiable causative process. Care is needed to prevent any secondary brain injury, which may include advanced respiratory and cardiovascular support. Monitoring is necessary to detect hypotension and hypoxia and steps taken to correct those conditions when recognized. Common complications may include traumatic injuries such as tongue lacerations or scalp lacerations . Convulsive status epileptic leads to brain damage on the cellular level and may itself be epileptogenic. Transformed or subtle generalized convulsive status epileptic or non convulsive seizures detected by EEG monitoring in critically ill patients may also contribute to brain laceration .

ELIGIBILITY:
Inclusion Criteria:

* Patient with recurrent attack of seizure and with prolonged seizure with prescribed treatment at home.
* Patients aged from 2 years to 18 years

Exclusion Criteria:

* First attack of seizure
* condition mimic epilepsy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric with seizure and take rescue intervention prehospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Aim of the study | Baseline
  1. Evaluation of prehospital rescue intervention of seizure management.
  2. To investigate the type of rescue medication,
     1. it's Efficacy.
     2. it's route of administration.
     3. Side effects of this drug.
     4. frequency .
     5. Indication of it's use.

SECONDARY OUTCOMES:
Seizure triggers | Baseline
  Seizures can be triggered by things in the environment. Seizure triggers don't cause epilepsy, but they may trigger seizures in people who have epilepsy.
  Most people with epilepsy don't have reliable triggers that always cause a seizure. However, they often can identify factors that make it easier to have a seizure. Possible :seizure triggers include
  * Illness
  * Skipping doses of antiseizure medicines or taking more than prescribed.
  * Dehydration
  * Lack of sleep
  * Flashing lights
  * Stress
  * Hormone changes during the menstrual cycle• Illicit drug use
  * Skipped meals

REFERENCES:
- [Background] Laccheo I, Sonmezturk H, Bhatt AB, Tomycz L, Shi Y, Ringel M, DiCarlo G, Harris D, Barwise J, Abou-Khalil B, Haas KF. Non-convulsive status epilepticus and non-convulsive seizures in neurological ICU patients. Neurocrit Care. 2015 Apr;22(2):202-11. doi: 10.1007/s12028-014-0070-0. PMID 25246236
- [Background] Silbergleit R, Durkalski V, Lowenstein D, Conwit R, Pancioli A, Palesch Y, Barsan W; NETT Investigators. Intramuscular versus intravenous therapy for prehospital status epilepticus. N Engl J Med. 2012 Feb 16;366(7):591-600. doi: 10.1056/NEJMoa1107494. PMID 22335736
- [Background] Cloyd J, Haut S, Carrazana E, Rabinowicz AL. Overcoming the challenges of developing an intranasal diazepam rescue therapy for the treatment of seizure clusters. Epilepsia. 2021 Apr;62(4):846-856. doi: 10.1111/epi.16847. Epub 2021 Feb 22. PMID 33617690
- [Background] Young GB, Claassen J. Nonconvulsive status epilepticus and brain damage: further evidence, more questions. Neurology. 2010 Aug 31;75(9):760-1. doi: 10.1212/WNL.0b013e3181f32141. No abstract available. PMID 20805520